CLINICAL TRIAL: NCT06913621
Title: The Use of High Bile-Binding Foods to Reduce Upper Gastrointestinal Bile Acid Concentrations: A Novel Intervention for Children at Risk for Aspiration-Associated Complications (Aim 3)
Brief Title: The Use of High Bile-Binding Foods to Reduce Upper Gastrointestinal Bile Acid Concentrations (Aim 3)
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel Rosen, Director, Aerodigestive Center, Boston Children's Hospital
Other Study IDs: IRB-P00049734 Aim 3
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-03

CONDITIONS: Feeding Difficulties; Gastrostomy; Aspiration
Keywords: blenderized; bile acid; gastrostomy; aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- amino acid-based formula
  Interventions: Drug: amino acid formula
- Low bile binding blenderized diet
  Interventions: Drug: low bile acid binding blenderized diet
- High bile binding blenderized diet
  Interventions: Drug: high bile acid binding blenderized diet

INTERVENTIONS:
Drug: amino acid formula — amino acid formula for 6 months
  Groups: amino acid-based formula
Drug: low bile acid binding blenderized diet — low bile acid binding blenderized diet for 6 months
  Groups: Low bile binding blenderized diet
Drug: high bile acid binding blenderized diet — high bile acid binding blenderized diet for 6 months
  Groups: High bile binding blenderized diet

SUMMARY:
Using a longitudinal cohort design, we will compare the impact of a high BA-binding blenderized diet compared to a low BA-binding blenderized diet and an amino acid-based formula, on gastrointestinal and pulmonary hospitalization and emergency room visit rates over six months.

ELIGIBILITY:
Inclusion Criteria:

* receive at least 80% of their nutritional needs via gastrostomy
* receive an International Dysphagia Diet Standardization Initiative level 4 commercial blend, home blend or amino acid-based formula
* receive their bolus feeds within 30 minutes or less.

Exclusion Criteria:

* have undergone anti-reflux surger
* receive post-pyloric feeds
* receive regular daily prophylactic antibiotics.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children requiring gastrostomy tube feeds for feeding difficulties
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
total hospitalization and emergency room visits rates | 6 months
  total hospitalization and emergency room visits rates between participants receiving H-BBB and those receiving L-BBB or an amino acid-based formula

SECONDARY OUTCOMES:
differences in pulmonary, gastrointestinal or ICU admission rates | 6 months
  differences in pulmonary, gastrointestinal or ICU admission rates between diets
differences in bile acid concentrations | 6 months
  differences in bile acid concentrations between diets
correlations between microbial abundance and diversity and hospitalization and emergency room visit rates | 6 months
  correlations between microbial abundance and diversity and hospitalization and emergency room visit rates
differences in metagenomic patterns between diets | 6 months
correlations between admission rates by diet type and short chain fatty acid concentrations | 6 months

IPD SHARING:
Plan to Share IPD: No